CLINICAL TRIAL: NCT04039321
Title: The Effect of Erector Spina Plane Block on Pulmonary Functions and Analgesic Consumption in Laparoscopic Sleeve Gastrectomy Surgery
Brief Title: Erector Spina Plane Block in Laparoscopic Sleeve Gastrectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Arzu Karaveli, study director, Antalya Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13/22
Record Dates: First submitted 2019-07-27; First posted 2019-07-31 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Obesity
Keywords: Erector spina plane block; Laparoscopic sleeve gastrectomy; Obesity; Postoperative pain; Pulmonary functions
MeSH Terms: conditions — Obesity; Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB group (Active Comparator): Before anaesthesia induction; bilateral ESP block will be performed under the guidance of USG. Patients will be administered paracetamol 1 gr IV every 8 hours in the postoperative period. If patients' NRS score will ≥4/10, 100 mg IV tramadol will be performed.
  Interventions: Drug: ESPB group
- Control group (Sham Comparator): Patients will be administered paracetamol 1 gr IV every 8 hours in the postoperative period. If patients' NRS score will ≥4/10, 100 mg IV tramadol will be performed.
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: ESPB group — USG probe will be placed in a longitudinal parasagittal orientation 3 cm lateral to T7 spinous process. The erector spinae muscles will be identified hyperechoic transverse process. The patient's skin will be anesthetized with 2% lidocaine. A 21-gauge 10-cm needle was inserted using an in-plane superior-to-inferior approach or an outplane approach. Following confirmation of the correct position of the needle with 5 ml normal saline, a dose of 20 ml %0.25 bupivacaine will be administered. The same procedure will be performed at the other site (totally 40 ml %0.25 bupivacaine). Standard pain follow up and monitorization will be performed.
  Arms: ESPB group
Drug: Control group — The patients in this group will be performed no block. Standard pain follow up and monitorization will be performed.
  Arms: Control group

SUMMARY:
The aim of the study is to evaluate the effect of erector spina plane (ESP) block on pulmonary functions and postoperative analgesic consumption in patients undergoing bariatric surgery.

DETAILED DESCRIPTION:
Optimal pain management is very important in obese patients. In the postoperative period, narcotic analgesics are often used to pain management. However, the use of narcotic analgesics in the postoperative period causes many undesirable adverse effects, especially sedation, dizziness, constipation, nausea, vomiting, muscle rigidity, tolerance, and respiratory depression.

The morbidly obese patients treated with narcotic analgesics increased risk for adverse effects such as atelectasis, hypoxemia, and postoperative ileus. Consequently, these are caused postoperative pulmonary complications, hypoxemia and longer lenght of hospital stay. Multimodal analgesia including local and regional anesthesia is recommended for morbidly obese patients.

In recent years, the ultrasound (USG) guided ESP block has been frequently used to eliminate postoperative pain and reduce narcotic analgesic use. In the literature, it has been shown that bilateral USG guided ESP block provides effective analgesia and decrease the analgesia requirements after laparoscopic cholecystectomy. Some case series and case reports has also been reported that ESP block provides effective analgesia after abdominal and bariatric surgeries.

The aim of the study is to evaluate the effect of erector spina plane (ESP) block on pulmonary functions and postoperative analgesic consumption in patients undergoing bariatric surgery. For this purpose, ASA II-III, patients over 18 years of age, BMI 40-60 kg/m2 and elective bariatric surgery planned patients will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) II-III
* 18-65 years
* body mass index (BMI) 40-60 kg/m2
* elective bariatric surgery

Exclusion Criteria:

* ASA ≥4
* under 18 years of age or over 65 years of age
* declining to give written informed consent
* have neurological and/or psychiatric disorders
* cooperation cannot be established
* accompanying laparoscopic cholecystectomy or paraumbilical hernia repair
* history of bariatric surgery
* the block cannot be applied due to bleeding disorders or localized skin infection at the injection site
* with hepatic, neuromuscular, cardiac and/or renal failure
* history of allergy to the local anesthetics
* patients undergoing open surgery
* patients with severe obstructive or restrictive lung disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
pulmonary function test | perioperative
  Pulmonary function test will be performed for all of them in the day before operation and 24 hours after the operation. Pulmonary function tests will assess via a portable spirometer with the patient in the sitting or semi-recumbent position.
analgesia consumption | 24 hours
  postoperative 24 hours

SECONDARY OUTCOMES:
Postoperative Numeric Rating Scale (NRS) score | postoperative 0, 1, 3, 6, 9, 12, 18, 24 hours
  postoperative pain assessment will be performed using NRS score (NRS 0=no pain, NRS 10= most severe possible). The NRS scores will be recorded at postoperative 0, 1, 3, 6, 9, 12, 18 and 24 hours
arterial blood gases | during the surgery
  intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Karaveli, Principal Investigator — Antalya TRH
Locations (1):
- Antalya Training and Research Hospital, Department of Anesthesiology and Reanimation, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chin KJ, Malhas L, Perlas A. The Erector Spinae Plane Block Provides Visceral Abdominal Analgesia in Bariatric Surgery: A Report of 3 Cases. Reg Anesth Pain Med. 2017 May/Jun;42(3):372-376. doi: 10.1097/AAP.0000000000000581. PMID 28272292
- [Background] Tulgar S, Kapakli MS, Senturk O, Selvi O, Serifsoy TE, Ozer Z. Evaluation of ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy: A prospective, randomized, controlled clinical trial. J Clin Anesth. 2018 Sep;49:101-106. doi: 10.1016/j.jclinane.2018.06.019. Epub 2018 Jun 15. PMID 29913392